CLINICAL TRIAL: NCT02896478
Title: Securing and Optimizing the Patient's Drug Therapy With Cancer: Clinical Pharmacy and Articulation With the City
Acronym: PRIMAC
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PRIMAC
Record Dates: First submitted 2016-08-31; First posted 2016-09-12 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2016-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention. Only observational study

SUMMARY:
The path of a patient depends largely on his health care network, that is to say of the interrelationships between health professionals who will be involved throughout his career. At the hospital, the transition points in the care process is a vulnerable time for the patient regarding the continuity of his medication. These transition points are the intake, the transfer and the outlet. In town, our health system must be able to build on the inter-city hospital, warranty essential guarantee of the continuity of care. However, there is often a breakdown in this relationship with more or less serious consequences ranging from simple dissatisfaction of the patient, to the realization of duplicate examinations or the use unjustified emergency and re-hospitalization. Medication errors can occur, resulting from incomplete information or poorly communicated in this city hospital interface.

The city hospital dysfunctions are mainly organizational, hospital being rather specialized therapeutic approach centered on pathology and medicine city instead focuses on a patient's overall approach.

The involvement of the pharmacist in the hospital, as the city is an interesting axis to develop. In town, the pharmaceutical nomadism, including in major cities remains low, patients generally have a dedicated pharmacies for the treatment of their serious or chronic pathologies. The development of the pharmaceutical folder today allows the pharmacies to access the history and the entire therapy of patients prescribed to town by different specialists and general practitioners, on the last 4 months. Its recent availability within our hospital Group allows us to consider its use to fully optimize the patient's drug monitoring.

DETAILED DESCRIPTION:
Hypothesis The involvement of hospital pharmacists from the admission of the patient in the oncology department until its release, with a comprehensive review of its treatment and anticipation of therapeutic needs when returning home and a joint organized with the community pharmacist and doctor, reduces the rate of drug discontinuity and thus improve its therapeutic management.

Goal

The investigators want to integrate and evaluate clinical pharmacist activities at different stages of the patient care process transition points:

* The admission by drug conciliation to determine exhaustively the medication history and the observed differences, and assess the patient's treatment adherence, to consider a revision of the treatment if necessary
* During the stay by daily pharmaceutical validation of drug prescriptions made in DxCare to play down the drug iatrogenic and participate in the definition of pharmacotherapy,
* In preparation for the release of the drug per patient reconciliation to inform and advise the patient about treatment and communicate relevant information to the city of health professionals.

  1. / DRUG RECONCILIATION TO ENTRY

     * Rational The investigators all remember, share different hospital functions, at least one example of Event Junk Medicated (EIM) suffered by a patient, the investigators participate in the management and from a medication error. The frequency of Adverse Event Graves (SAEs) exclusively related to health products is estimated at 1.7 per 1000 SAE avoidable hospital days, or just over 1 SAEs per day for a 1,000 bed hospital. This study showed a stronger exposure to preventable SAEs among elderly and vulnerable. Indeed, promoting factors the occurrence of iatrogenic injuries for this population are manifold: multi-pathologies, polypharmacy, organic impairment, cognitive impairment, inadequate mode of administration. Some of these therapeutic errors are the result of poor communication between the city and the hospital, leading to hospitalized patients for whom took home treatments are not exhaustively known. It is also estimated that 67% of drug history of patients have one or more medication errors and that 46% of these errors occur at the time of the drafting of a new order to the entrance or exit of the patient 's hospital. The EQUIP study showed that the risk of prescription errors was increased by 70% during the intake phase of the patient from the hospital phase. On the other hand, it has been reported that 60% of cancer patients use complementary and alternative medicine, for which we must be vigilant about taking these medications potentially iatrogenic (MAC-AERIO study 2010).

Goal Detect differences in prescription between the city and the hospital in establishing a complete and exhaustive list of treatments taken by the patient before hospitalization, avoiding medication errors, appearance starting point EIG.

procedure The hospitalization of Medical Oncology Service has 20 beds (14 traditional hospital beds and six weeks of hospital beds) with an average rate of entries per day of 3-4 patients, 1 to 2 per week are new patients. Patients will be seen by a hospital pharmacist within <24h of admission, or <72 h during late entry on Friday, Saturday, and Sunday morning.

1. / The reconciliation begins with a review of treatments called Bilan Medicated Optimized (BMO). The list to be drawn regarding medications taken by the patient whether prescribed or not. To formalize, it is necessary to conduct an interview with the patient and / or his entourage as well as city health professionals or other care facilities if any. The first source of information is that we will exploit the patient's pharmaceutical record (if open), accessible via its vital card and resuming treatment provided during the last 4 months. If drugs are brought home by the patient, they are another useful source of information. BMO This will be achieved in 2 ways:

   * Proactive Patient entering Sunday to Thursday. The drafting of the first order in the service has not yet taken place, BMO is then used to prescriber for the drafting of the Ordinance for Medicinal Products for admission (OMA). Accordingly, the error of drug therapy is intercepted before it takes place. This option requires that conciliation by the pharmacist is made early in the patient's care in the hospital.
   * Retroactive for patients who already have a prescription in hospital © DxCare following their admission. BMO is established after drafting the OMA. It can then be discrepancies that conciliation will allow to intercept and correct. It follows writing additional information or a new prescription to correct the detected differences.
2. / The differences observed may be unintentional (medication errors) and correspond to involuntary treatment changes and are likely to generate an adverse event for the patient, or intentional but not documented and correspond to voluntary changes in treatment, the reasons are not indicated in the patient file. It may be an addition, modification or interruption of a medicament. This lack of information is likely to generate a medication error later. The characterization of the differences will result in 3 steps:

   * Each drug line is characterized by medical decision that seems to have been taken. The drug is thus considered stopped, suspended, continued in the state, continued with amendment, substituted or added.
   * Then the search of the annotated medical decision in the patient's file shows that if the decision is documented or not. When it is, the treatment line is validated. When it is not, it is concluded that there was a discrepancy.
   * At this late stage, the physician participation is mandatory to describe the degree of intent of the undocumented divergence: divergence is characterized as intentional or unintentional. Following the implementation of the reconciliation rule, three decisions are possible for each drug line studied:
   * The drug is validated online
   * In case of undocumented intentional discrepancy, the medical decision is to explain by filling in the patient file
   * In case of unintended discrepancy, the prescription is correct, there is a medication error. Any deviation must be documented at BMO. The lack of information can leave wrong to think that this discrepancy is intentional or not, hence the importance of documenting prescription for medical decision is explicit. By cons, a gap that is properly called unintentional must be corrected: it is a drug error can cause harm to the patient if it is not caught.
3. / The finalized conciliation document is then validated by the hospital pharmacist and ends up embedded in the patient record to be reused during a transfer or discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patient accepting to be roll on

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted in oncology unit at Paris Saint joseph Hospital
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Assessment of change of the Number of pharmaceutical consultations | Day 0, Day 3, day 30
Assessment of change of the Number of patients discharged | Day 0, Day 3, day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided